CLINICAL TRIAL: NCT02141386
Title: Plasticity-based, Adaptive, Computerized Cognitive Remediation Treatment (PACR) for Adults With Multiple Sclerosis (MS)
Brief Title: Computerized Cognitive Exercise Training Treatment for Adults With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stony Brook University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Lauren Krupp, Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG4808A81
Record Dates: First submitted 2014-02-14; First posted 2014-05-19 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cognitive remediation; Plasticity-based, adaptive, computerized cognitive remediation; Cognitive impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Treatment A (Experimental): plasticity-based, adaptive, computerized cognitive remediation (PACR)
  Interventions: Other: PACR (Plasticity-based, Adaptive, Computerized Cognitive Remediation)
- Treatment B (Active Comparator): Ordinary Computer Games (an "active control condition")
  Interventions: Other: PACR (Plasticity-based, Adaptive, Computerized Cognitive Remediation)

INTERVENTIONS:
Other: PACR (Plasticity-based, Adaptive, Computerized Cognitive Remediation)

SUMMARY:
Cognitive impairment remains a major disability for individuals with multiple sclerosis (MS). The primary objective of this study is to evaluate the efficacy for treating MS-associated cognitive deficits using a unique computer-based plasticity-based and adaptive cognitive remediation treatment (PACR) compared to a computer-based control. This novel cognitive remediation approach has led to striking improvements in cognitive functioning in other disorders (schizophrenia, traumatic brain injury, aging, and dementia) but has never been applied to individuals with MS. The investigators will enroll 136 MS participants who will be randomized in a 2:1 pattern to complete either the treatment or control condition for 60 hours across a 12-week treatment period. Both the treatment and control conditions will be accessed remotely by the subjects from a study-provided laptop computer. Study outcomes will include program compliance, performance on study tasks and neuropsychological measures, quality of life and functional status. Given the success of this program with other disorders and strong preliminary data from our feasibility study, the investigators believe PACR is an exciting untapped opportunity to improve cognition in individuals with MS.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Definite MS Diagnosis, any subtype [83]
* Probable cognitive impairment as defined by a score ≤ 1 SD below the mean of normative data on the SDMT
* Concurrent medications to be kept constant over three months (as possible)
* No relapse or steroids in previous month
* Reading score on WRAT-3 of 37 or greater
* Visual, auditory and motor capacity to operate computer software, as judged by treating neurologist or study staff
* Willing to sign Agreement to Borrow Laptop

Exclusion Criteria:

* History of mental retardation, pervasive developmental disorder or other neurological condition associated with cognitive impairment
* Primary psychiatric disorder that would influence ability to participate
* Other serious uncontrolled medical condition (e.g., cancer or acute myocardial infarction)
* Alcohol or other substance use disorder
* History of computer-based training manufactured by Posit Science
* Learned English language after 12 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
A composite derived from a standardized battery of neuropsychological tests | 12weeks
  Covariates will include baseline cognitive status, PACR program compliance, PACR task improvement, and participant-reported outcomes

SECONDARY OUTCOMES:
A timed measure based on direct observation of functional performance | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

REFERENCES:
- [Derived] Charvet LE, Yang J, Shaw MT, Sherman K, Haider L, Xu J, Krupp LB. Cognitive function in multiple sclerosis improves with telerehabilitation: Results from a randomized controlled trial. PLoS One. 2017 May 11;12(5):e0177177. doi: 10.1371/journal.pone.0177177. eCollection 2017. PMID 28493924